CLINICAL TRIAL: NCT06552949
Title: Prospective Cohort Study on Emergent Laparoscopic Cholecystectomy Guided by Indocyanine Green (ICG) Fluorescence Versus Conventional Laparoscopic Operation
Brief Title: A Prospective Cohort of Emergent Laparoscopic Cholecystectomy in PUMCH
Acronym: ELC-PUMCH
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiaofei Liu, Clinical Associate professor, Peking Union Medical College Hospital
Other Study IDs: K6454-K24C2458
Record Dates: First submitted 2024-08-06; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Acute Cholecystitis
Keywords: Emergent laparscopic cholecystectomy; indocyanine green fluorescence; surgical outcome; economic effectiveness; acute cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patient undergoing emergent laparoscpic cholecystectomy guided by indocyanine green cholangiography (ELC-ICGC)
  Interventions: Procedure: Emergent laparoscopic cholecystectomy guided by ICG cholangiography (ELC-ICGC)
- Control group: Patient undergoing emergent conventional laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Emergent laparoscopic cholecystectomy guided by ICG cholangiography (ELC-ICGC) — Emergent conventional laparoscopic cholecystectomy
  Groups: Study group

SUMMARY:
A prospective cohort study comparing the surgical outcome of patients who underwent emergent laparoscopic cholecystectomy guided by indocyanine green cholangiography (ELC-ICGC) versus conventional laparoscopic operation. The patients were recruited in the Peking Union Medical Colleg Hospital emergency department from 1st August 2020 to 1st Feburary 2024. A database was prospectively established to collect related data. The surgical outcomes of ELC-ICGC and conventional ElC will be compared.

DETAILED DESCRIPTION:
Acute calculous cholecystitis, typically occurs in patients with gallstones, accounts for 90 to 95% of acute cholecystitis. Emergent laparoscopic cholecystectomy (ELC) is the major treatment option. Traditionally, the time frame for ELC is generally considered to be within 72 hours from the onset of symptoms. However, with the development of surgical techniques, nowadays, ELC is also considered for patients with symptoms onset within 10 days and hospital stays within 7 days. The determination of the time frame for ELC in acute cholecystitis is primarily based on the risk of complications occurring. Comparing to delayed laparoscopic cholecystectomy (DLC), ELC has advantages in post-operative complications in patients with symptoms onset within 72 hours. Post-operative complications for both DLC and ELC include bile leaks, intestinal obstruction, ascites, intraperitoneal hemorrhage, would bleeding and hematoma, wound infection and calculus remaining. Most of them associate with intraoperative procedures. Emergent laparoscopic cholecystectomy guided by indocyanine green (ICG) cholangiography (ELC-ICGC), comparing to conventional LC, potentially can help the surgeons to identify bile tracts and therefore may reduce the complications.

From August 1st 2020, the AC patients undergoing LC in PUMCH were prospecteively registered and a database was established to collect related data.

Till 1st Feburary 2024, about 750 cases of ELC were performed. The surgeons chose to perform either conventional ELC or ELC-ICGC based on their discretion. The patients were followed up within one month after discharge in out patient clinic or telephone interview. We plan to analyze the data from the prospectively established- database.

The surgical outcomes are evaluated by both intraoperative events and postoperative events. Intraoperative events contain the following items: (1) incidence of intraoperative accidental bile tract injury, (2) intraoperative bleeding (volume), (3) operation time. Postoperative events contain the following items: (1) incidence of complications staging 2 and above according to Clavien Dindo Grade during hospital stay, (2) duration of postoperative hospital stay. The economic effectiveness is evaluated by cost of hospital stay.

The surgical outcomes of these two procedures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent ELC performed by the emergent surgeon team Approval to participate

Exclusion Criteria:

* Patients with incomplete medical records. Patients have other emergent conditions which warrant other emergent operations or major treatment simultaneously besides ELC.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All of the hospitalized patients who underwent ELC by the emergent surgery team from August 1st 2020 to 1st Feburary 2024 in the Department of Emergency in Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
incidence of intraoperative accidental bile tract injury | within 1 month
  The primary outcome is incidence of intraoperative accidental injury involving the bile tract in emergent laparscopic cholecystectomy (ELC) guided by ICG fluorescence. The injury manifests as biliary obstruction, biliary leak, or biliary stricture. Medical records will be reviewed to identify an intraoperative bile tract injury event. Incidence of intraoperative accidental bile tract injury will be collected and comparison between study group (ELC guided by ICG fluorescence) and control group (conventional ELC) will be made
incidence of complications | within 1 month
  incidence of complications staging 2 and above according to Clavien Dindo Grade during hospital stay

SECONDARY OUTCOMES:
intraoperative bleeding (volume) | Intraoperative
  Volume of intraoperative bleeding during the operation
duration of postoperative hospital stay | within 1 month
  Days of postoperative hospital stay
total medical expense | within 1 month
  Cost during hospital stay
operation time | Intraoperative
  from cutting the incison to ending the suturing of the incision

CONTACTS AND LOCATIONS:
Overall Officials: Qiaofei Liu, M.D, Study Chair — Department of General Surgery, Peking Union Medical College Hospital
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Peking Union Medical College & Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No